CLINICAL TRIAL: NCT07122648
Title: A Prospective, Multi-center, Randomized, Double-blinded, Placebo-controlled, Parallel, Phase 2 Trial to Evaluate the Efficacy, Safety of PN-101(Mitochondria Isolated From Allogeneic Umbilical Cord-derived Mesenchymal Stem Cells) Single Dose in Patients With Refractory Polymyositis or Dermatomyositis
Brief Title: Phase 2 Trial to Evaluate the Efficacy, Safety of Allogeneic Mitochondria (PN-101) in Patients With Refractory Polymyositis or Dermatomyositis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paean Biotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN-101-201
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: mitochondria
MeSH Terms: conditions — Polymyositis; Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator)
  Interventions: Biological: placebo
- 300 ug of PN-101 group (Experimental)
  Interventions: Biological: PN-101
- 600 ug of PN-101 group (Experimental)
  Interventions: Biological: PN-101

INTERVENTIONS:
Biological: placebo — Participants will receive a single IV dose of 300 µg of placebo
  Arms: Placebo Group
Biological: PN-101 — Participants will receive a single IV dose of 300 µg of PN-101
  Arms: 300 ug of PN-101 group
Biological: PN-101 — Participants will receive a single IV dose of 600 µg of PN-101.
  Arms: 600 ug of PN-101 group

SUMMARY:
The efficacy of PN-101 in subjects with polymyositis or dermatomyositis will be evaluated at Week 12 using IMACS-TIS in comparison with the placebo control group. The safety and efficacy will be evaluated following administration of PN-101 to subjects with polymyositis or dermatomyositis, in comparison with the placebo group

DETAILED DESCRIPTION:
This Phase II clinical trial involves patients diagnosed with polymyositis or dermatomyositis.

* Only subjects who have voluntarily provided written informed consent and have been determined to meet the inclusion/exclusion criteria will participate in this clinical trial.
* Subjects will be randomly assigned in a 1:1:1 ratio to the PN-101 300 ug group, 600 ug group, or placebo control group according to their randomization number, and stratified based on the diagnosis of either polymyositis or dermatomyositis.
* The investigator will administer a single intravenous dose of either the placebo or the investigational product to subjects in the placebo control group and the treatment groups.
* Each subject who receives the investigational product will be monitored for any acute adverse events, such as hypersensitivity, within 30 minutes after administration.
* Safety and efficacy will be evaluated according to the visit schedule after administration of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 19 years or more
2. A subject who is diagnosed with polymyositis or dermatomyositis and satisfies all of the followings:

   * Clinical profile: Slowly progressing clinical profile with symmetrical and apparent muscular weakness confirmed at the proximal muscle (in case of dermatomyositis, clinical findings related with characteristic skin symptoms*)

     * Gottron's papules or sign, erythema purpura, poikiloderma, calcinosis cutis, etc.
   * Serum test: Serum creatine kinase (CK) elevated (CK ≥ 1.3 × upper limit of normal (ULN)) or serum myositis-specific antibodies (MSA) positive
   * Electromyography (EMG): Presence of a finding that indicates myopathy
3. Baseline (prior to the investigational product administration) manual muscle testing-8 (MMT-8) result < 125/150 (bilaterally), and at least 2 of the following International Myositis and Clinical Studies Group (IMACS) core set results

   * Physician global disease activity [visual analogue scale (VAS)] ≥ 2 cm
   * Patient global disease activity [VAS] ≥ 2 cm
   * Health assessment questionnaire (HAQ) disability assessment ≥ 0.25
   * 1 or more items with the serum muscle enzyme > 1.3 × ULN
   * Global extramuscular disease activity [VAS] > 1 cm
4. Individuals who are currently receiving glucocorticosteroids and/or steroid-sparing drugs such as immunosuppressants or immunomodulators for the treatment of polymyositis or dermatomyositis but are deemed to have an inadequate response to treatment, or who are unable to continue existing treatment due to drug-related adverse events or side effects (however, during the clinical trial, the dosage of steroids and immunosuppressants may be adjusted within 20% of the dose prior to the study participation)
5. Individuals who are receiving exercise or physical therapy and have agreed to maintain the same intensity and frequency of their current therapy
6. A subject who fully understands the trial and provided voluntary written consent to take part in the trial

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible to participate in this clinical trial:

1. A subject with clear muscular damage, with the VAS-based myositis damage index (MDI) of ≥ 5 at screening
2. A subject with the following medical history or surgical history

   * A surgical operation history within 12 weeks of screening
   * Malignant tumor within 5 years of screening (excluding a subject who passed 3 years or more from complete recovery of cervical cancer or skin squamous cell carcinoma)
3. Patients diagnosed with polymyositis or dermatomyositis before the age of 10 (Juvenile PM or Juvenile DM)
4. A patient with severe respiratory muscular weakening or interstitial pulmonary disease (a patient who has no moderate or severe dyspnea and has stable interstitial pneumonia may participate)
5. A patient with the following comorbidity at screening

   * Acute viral infection or severe infection
   * Active hepatitis B (e.g.: HBsAg positive and HBV DNA detected) or hepatitis C (e.g.: Anti-HCV positive and HCV RNA [qualitatively] detective)
   * Human Immunodeficiency virus (HIV) positive
   * Findings of muscular inflammation or myopathy other than the indication (inclusion body myositis (IBM), drug-induced myopathy, amyloid myopathy, myotonic dystrophy, etc.)
   * Autoimmune disease such as rheumatoid arthritis (RA), systemic lupus erythematosus, psoriatic arthritis, etc. (however, in case of the overlap syndrome, a subject may participate if diseases other than inflammatory myositis are stable and myositis is thought to be due to inflammatory myositis.)
   * Findings of cardiac disorder such as moderate or severe heart failure (New York Heart Association Class III/IV) or QT corrected interval prolonged
   * Serious disease that may affect this study, at the discretion of the investigator (neurological disorder, cardiovascular disorder, uncontrolled blood pressure or diabetes, etc.)
6. Hematological, renal and hepatic dysfunction based on the following laboratory findings at screening

   * Glomerular filtration rate (GFR)* < 45 mL/min *eGFR (mL/min/1.73m^2) = 175 × (serum creatinine concentration (mg/dL))^-1.154 × (age)^-0.203 × (0.742 in female) [modification of diet in renal disease (MDRD) formula]
   * Hemoglobin < 10 g/dL
   * White blood cell (WBC) count < 3.0×10^9/L
   * Absolute neutrophil count (ANC) < 1.5×10^9/L (1500/mm^3)
   * Platelet count < 100×10^9/L
   * AST and ALT > 2.5 × ULN (except for the elevation due to muscle enzyme at the discretion of the investigator)
   * Alkaline phosphatase (ALP) > 2.5 × ULN
   * Total bilirubin > 1.5 × ULN (> 3 × ULN, in case of Gilbert's syndrome)
   * Thyroid stimulating hormone level exceeding the normal range (however, if the level exceeds the normal range due to the study indication at the discretion of the investigator, the subjects are allowed to enroll.)
7. A subject with a difficulty in the efficacy assessment including the muscular strength assessment during the trial
8. A subject who is determined to require prohibited concomitant treatment during the trial
9. Pregnant woman and lactating mother or woman of childbearing potential and man who is planning to have a child or not willing to practice acceptable contraception* for 36 weeks after the last dosing date *Hormonal contraception, intrauterine device or intrauterine system implant, surgical sterilization procedure/operation (vasectomy, tubal ligation, etc.)
10. Participation in other clinical trial and administration of an investigational product or application of an investigational device within 4 weeks or half-life x 5 (whichever is longer) prior to screening
11. A subject who is otherwise ineligible for this trial, at the discretion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
International Myositis And Clinical Studies group-Total Improvement Score (IMACS-TIS) | 12 weeks after the IP administration
  Assessment of IMACS-TIS at Week 12 (Visit 6) after the IP administration. Total Improvement Score (TIS) based on absolute percentage change is assessed scale 0 to 100. Higher score indicates greater improvement.

SECONDARY OUTCOMES:
International Myositis And Clinical Studies group-Total Improvement Score (IMACS-TIS) | 4 weeks, 8 weeks , and 16 weeks after the IP administration
  Assessment of IMACS-TIS at week 4, week 8, and week 16 after the IP administration. Total Improvement Score (TIS) based on absolute percentage change is assessed scale 0 to 100. Higher score indicates greater improvement.
Response rate of IMACS-TIS | 4 weeks, 8 weeks , 12 weeks, and 16 weeks after the IP administration
  Proportion of subjects with the IMACS-TIS ≥ 20 at week 4, week 8, week 12, and week 16 after IP administration
Changes of Core Set Activity Measures(CSAM) | Visit 2(Day 1), Visit 4(4 weeks), Visit 5(8 weeks), Visit 6(12 weeks), Visit 7(16 weeks)
  Changes in CSAM for the IMACS assessed at week 4, week 8, week 12, and week16 after the IP administration from the baseline (Visit 2). The core set for the IMCS consists of six components: physician global disease activity, patient global disease activity, MMT-8, extramuscular activity, HAQ, and serum muscle enzyme levels.
Changes of Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) | Visit 2(Day 1), Visit 4(4 weeks), Visit 5(8 weeks), Visit 6(12 weeks), Visit 7(16 weeks)
  Changes in CDASI assessed at week 4, week 8, week 12 and week 16 after the IP administration from the baseline (Visit 2) for dermatomyositis only.
Changes of Peak Pruritus Numeral Rating Scale(PPNRS) | Visit 2(Day 1), Visit 4(4 weeks), Visit 5(8 weeks), Visit 6(12 weeks), Visit 7(16 weeks)
  Changes in PPNRS assessed at week 4, week 8, week 12 and week 16 after the IP administration from the baseline (Visit 2) for dermatomyositis only. The intensity of pruritis is assessed on a patient reported scale 0 to 10.

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Chung-Ang University Gwang Myeong Hospital, Gwangmyeong, Gyeonggi-do
  - Kyung Hee University Medical Center, Seoul
  - Seoul National University, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No